CLINICAL TRIAL: NCT03425071
Title: Monitoring Intracellular Concentration and Pharmacodynamic Effects of Tacrolimus in Peripheral Blood T CD4+ and B CD19+ Lymphocytes of Kidney Transplant Recipients
Brief Title: Monitoring Concentration and Pharmacodynamic Effects of Tacrolimus in Peripheral Blood Lymphocytes of Kidney Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Maria da Luz Fernandes (Unknown); Paschoalina Romano (Unknown); Persio de Almeida Rezende Ebner (Unknown); Nairo Massakazu Sumita (Unknown); Veronica Porto Carreiro de Vasconcelos Coelho (Unknown); Fabiana Agena (Unknown); Elias David Neto (Unknown); Nelson Zocoler Galante (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAAE 41558915900000068
Record Dates: First submitted 2018-01-30; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Kidney Transplantation; Rejection
Keywords: Tacrolimus; T Lymphocytes; B lymphocytes; Monitoring, Immunologic
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Healthy volunteers - subjects without exposure to tacrolimus. Blood samples from these subjects will be used in "in vitro" experiments.
- kidney transplant (KTx) months 1-2: Kidney transplant recipients recruited during the months 1 to 2 of follow up after kidney transplantation surgery. These are subjects expected to be exposed to high blood levels of tacrolimus. Blood samples from these subjects will be used in "ex vivo" experiments.
- KTx months 4-5: Kidney transplant recipients recruited during the months 4 to 5 of follow up after kidney transplantation surgery. These are subjects expected to be exposed to standard blood levels of tacrolimus. Blood samples from these subjects will be used in "ex vivo" experiments.

SUMMARY:
Therapeutic drug monitoring (TDM) of immunosuppressive drugs is used to improve the immunosuppressive effect while minimizing the toxicity related to exposition to high serum levels. Although TDM is widely used in clinical practice, a significant number of kidney transplant recipients have acute allograft rejection in the first year after transplantation. To improve the use of immunosuppressive drugs, new approaches of TDM have been developed. Monitoring drug concentrations at lymphocytes of peripheral blood is considering promising because it indicates the availability of the drug directly in the target sites of immunosuppression. The present study intends to establish the concentration profile of tacrolimus in the peripheral blood in parallel with the concentration profile inside T and B lymphocytes of peripheral blood of kidney transplant recipients, and correlates them with the expected pharmacological effects. The pharmacological effects of tacrolimus in calcineurin dependent and calcineurin independent (mitogen-activated protein kinase (MAPK) dependent) activation pathways will be assessed by measuring activated nuclear factor of activated T cells (NFAT) and p38, respectively, by flow cytometry. The expression of interleukin (IL) - 2 and IL-10 by T and B lymphocytes, respectively, will be also used to monitoring the pharmacodynamic effects of tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients with a well functioning graft (serum creatinine ≤ 2,0 mg/dL at inclusion)
* Must be on tacrolimus therapy
* Must be on short term follow up time (1 to 5 months) after surgery

Exclusion Criteria:

* A concomitant second solid organ transplant
* Immunosuppression not containing tacrolimus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will include kidney transplant recipients followed at Hospital das Clínicas da Faculdade de Medicina da USP.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between blood and intracellular levels of tacrolimus | From 1 up to 5 months post transplantation
  The concentration of tacrolimus will be determined in the whole blood, in T CD4+ cell suspension and in B CD19+ cell suspension prepared from one blood sample per patient subject. The correlations among concentrations of tacrolimus in the 3 different cell matrices will be established.

SECONDARY OUTCOMES:
Correlation among intracellular levels of tacrolimus and its pharmacological effects | From 1 up to 5 months post transplantation
  The pharmacological effects of tacrolimus will be measured as the inhibition of the nuclear translocation of NFAT transcription factor, the phosphorylation state of p38 MAP kinase and the production of interleukin 2 and 10 by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Z Galante, PhD, Principal Investigator — Kidney Transplantation Service - University of Sao Paulo
Locations (1):
- Hospital das Clínicas - University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Romano P, da Luz Fernandes M, de Almeida Rezende Ebner P, Duarte de Oliveira N, Mitsue Okuda L, Agena F, Mendes ME, Massakazu Sumita N, Coelho V, David-Neto E, Zocoler Galante N. UPLC-MS/MS assay validation for tacrolimus quantitative determination in peripheral blood T CD4+ and B CD19+ lymphocytes. J Pharm Biomed Anal. 2018 Apr 15;152:306-314. doi: 10.1016/j.jpba.2018.01.002. Epub 2018 Jan 5. PMID 29471254